CLINICAL TRIAL: NCT02181920
Title: Analgesic Effect of a New Metamizol Oral Pharmaceutical Form for the Treatment of the Neoplastic Chronic Pain: Randomized, Double-blind Crossover Clinical Trial Between Metamizol, Diclofenac and Placebo
Brief Title: Metamizol for the Treatment of Neoplastic Chronic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1093.14
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dipyrone; Diclofenac

ARMS (4):
- Metamizole - Diclofenac (Experimental): metamizole followed by diclofenac
  Interventions: Drug: Metamizole; Drug: Diclofenac; Drug: Diclofenac placebo; Drug: Metamizole placebo
- Diclofenac - Metamizole (Experimental): diclofenac followed by metamizole
  Interventions: Drug: Metamizole; Drug: Diclofenac; Drug: Diclofenac placebo; Drug: Metamizole placebo
- Metamizole - Placebo (Experimental): metamizole followed by placebo
  Interventions: Drug: Metamizole; Drug: Diclofenac placebo; Drug: Metamizole placebo
- Placebo - Metamizole (Experimental): placebo followed by metamizole
  Interventions: Drug: Metamizole; Drug: Diclofenac placebo; Drug: Metamizole placebo

INTERVENTIONS:
Drug: Metamizole
Drug: Diclofenac
  Arms: Diclofenac - Metamizole; Metamizole - Diclofenac
Drug: Diclofenac placebo
Drug: Metamizole placebo

SUMMARY:
Study to evaluate the efficacy of metamizole in reducing morphine requirements in patients with moderate to severe chronic cancer pain in comparison to administration of placebo or diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with neoplastic chronic pain requiring morphine treatment

Exclusion Criteria:

* Karnofsky index less than 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2000-03; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Change in morphine requirement | Baseline, 9 days